CLINICAL TRIAL: NCT04105634
Title: Molecular Imaging of the Underlying Mechanism of Cardiotoxicity in Patients With Cardiac Amyloidosis Using Positron Emission Tomography (PET/CT)
Brief Title: Molecular Imaging of the Underlying Mechanism of Cardiotoxicity in Patients With Light Chain Amyloidosis Using PET/CT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833485
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inflammation group (Experimental): Patient diagnosed with Cardiac Amyloidosis
  Interventions: Drug: FNOS
- Amyloid group (Experimental): Patient diagnosed with Cardiac Amyloidosis
  Interventions: Drug: Florbetaben

INTERVENTIONS:
Drug: FNOS — The imaging drug used for this group is called 18F-NOS, it is an experimental imaging drug that has not yet been approved by the Food and Drug Administration (FDA) for use except in a research study. Subject will not receive the results or feedback from the study participation, the images may be reviewed with subject or her/his doctor upon request but will not be used to make decisions about subject medical care.
  Other Names: [18F]-6-(2-fluoro-propyl)-4-methylpyridin-2-amine
  Arms: Inflammation group
Drug: Florbetaben — The imaging drug used for this group is called Florbetaben, it is an FDA approved radioactive PET tracer used to image amyloid plaques in the body. Although not yet FDA approved for this purpose, it has already been used clinically to image amyloid in other parts of the body. Subject will not receive the results or feedback from the study participation, the images may be reviewed with subject or her/his doctor upon request but will not be used to make decisions about subject medical care.
  Other Names: Neuraceq
  Arms: Amyloid group

SUMMARY:
The research study is being conducted to test how two different types of Positron Emission Tomography (PET/CT) scans could be used to image a type of heart disorder called amyloidosis (AL). There will be two groups in the study. One group will have PET/CT scans using an imaging drug called 18F-NOS and the other group will have PET/CT scans using a drug called Florbetaben. subject will be assigned to one of the groups when she/he agrees to be in the study.

DETAILED DESCRIPTION:
Immunoglobulin light chain (LC) amyloidosis (AL) is an underdiagnosed monoclonal plasma cell proliferative disorder caused by extracellular deposition of AL fibrils in various tissues and organs, causing disease by progressively damaging the structure and function of the affected tissue/organ. The heart is the most commonly involved organ (~75%),9 and the extent and severity of cardiac involvement continue to be the main limitation for successful treatment. Although it remains high, the 6-month mortality rate has improved significantly over the last decade (24% vs. 37%; P<0.001) due to earlier diagnosis, better treatment options, and the advent of sensitive serologic biomarkers to assess for early treatment response,10 in particular serum free light chains (FLC), which permit the differentiation of patients who achieve complete response (CR) and very good partial response (VGPR) from those with partial or no response. N-terminal fragment of the pro-brain natriuretic peptide (NT-proBNP) has also become a key biomarker for detection and risk-stratification of patients with cardiac AL amyloidosis, and is now routinely employed in clinical trials as a surrogate end point for survival. A large retrospective landmark analysis established that achievement of a CR or VGPR at 6 months post-initiation of therapy, or achievement of an NTproBNP response 6 months post-initiation of therapy, defined as a 30% reduction and absolute reduction ≥ 300 pg/mL from baseline for subjects with baseline levels ≥ 650 pg/mL, was strongly associated with improved overall survival (insert Palladini et al, JCO 2012).

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be at least 18 years of age
2. Have an established diagnosis of AL amyloidosis based on standard criteria and planning to start systemic therapy.
3. Have cardiac involvement as defined by all of the following:

   * Past documented or presently noted clinical signs and symptoms supportive of a diagnosis of heart failure in the setting of a confirmed diagnosis of AL amyloidosis in the absence of an alternative explanation for heart failure
   * Either an endomyocardial biopsy demonstrating AL amyloidosis or an echocardiogram demonstrating a mean left ventricular wall thickness at diastole >12mm in the absence of other causes (e.g. severe hypertension, aortic stenosis), which would adequately explain the degree of wall thickening
   * NT-proBNP ≥ 650 pg/mL
4. Participants should fall into 1 of the following 2 categories:

   1. Treatment-naïve or have completed no more than 1 cycle of initial therapy, OR
   2. Relapsed after 1 or more prior therapies, and at least 6 months from last treatment
5. Have serum free light chain (FLC) differential (defined as amyloid-forming FLC minus non-amyloid-forming FLC) ≥ 50 mg/L.
6. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast feeding at the time of the PET/CT scan will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential before the injection of radiotracer.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
4. Less than 6 months life expectancy as deemed by a treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Measure uptake of [18F]NOS and Florbetaben in patients with AL before and ~4 months (2 +/- weeks) after starting standard therapy using PET/CT | 4 months
  Measure uptake of [18F]NOS and Florbetaben in patients with AL before and ~4 months (2 +/- weeks) after starting standard therapy and describe the distributions of uptake values at each time point. Compute post-/pre-treatment fold change in [18F]NOS and Florbetaben uptake and describe its distribution.

SECONDARY OUTCOMES:
Describe fold changes in [18F]NOS uptake in patients who have a complete response or very good partial response vs patients who have a partial or no response to therapy at ~4 months. | 4 months
  Describe fold changes in [18F]NOS uptake in patients who have a complete response or very good partial response vs patients who have a partial or no response to therapy at ~4 months.
Describe fold changes in [18F]NOS uptake in patients who have an NT-proBNP response at ~4 months vs patients who have no response or progression | 4 months
  Describe fold changes in [18F]NOS uptake in patients who have an NT-proBNP response at ~4 months vs patients who have no response or progression
Describe fold changes in Florbetaben uptake in patients who have an NT-proBNP response at ~4 months vs patients who have no response or progression | 4 months
  Describe fold changes in Florbetaben uptake in patients who have an NT-proBNP response at ~4 months vs patients who have no response or progression

CONTACTS AND LOCATIONS:
Overall Officials: Paco Bravo, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States